CLINICAL TRIAL: NCT06806176
Title: Effectiveness and Acceptability of Cognitive Analytic Therapy Guided Self-help (CAT-GSH) for Anxiety and Depression for Returning Patients in NHS Talking Therapies Services
Brief Title: Effectiveness of CAT-GSH for Returning Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: Catalyse CAT Limited (Unknown); Tameside and Glossop Talking Therapies service (Unknown); Leeds Mental Wellbeing service (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 191606
Record Dates: First submitted 2025-01-31; First posted 2025-02-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-01

CONDITIONS: Anxiety; Depression
Keywords: Cognitive analytic therapy (CAT); Guided self-help; NHS Talking Therapies; returning patients; Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Participants will have a choice between CBT guided self-help and CAT guided self-help.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-GSH arm (Active Comparator): CBT-GSH group
  Interventions: Behavioral: Cognitive behavioural therapy guided self-help (CBT-GSH)
- CAT-GSH arm (Active Comparator): CAT-GSH group
  Interventions: Behavioral: Cognitive analytic therapy guided self-help (CAT-GSH)

INTERVENTIONS:
Behavioral: Cognitive analytic therapy guided self-help (CAT-GSH) — Six session CAT-GSH treatment
  Arms: CAT-GSH arm
Behavioral: Cognitive behavioural therapy guided self-help (CBT-GSH) — Six session CBT-GSH treatment
  Arms: CBT-GSH arm

SUMMARY:
The goal of this clinical trial is to learn if cognitive analytic therapy-guided self-help (CAT-GSH) is comparable to cognitive behavioural therapy-guided self-help (CBT-GSH) in terms of whether it is effective and acceptable for people with anxiety or low mood, who are returning to NHS Talking Therapy services for further treatment. The main questions it aims to answer are:

* Does CAT-GSH work well and feel acceptable for people coming back to the Talking Therapies service, compared to CBT-GSH, when taking their characteristics (like age) into account
* Does CAT-GSH work well and feel acceptable for people coming back to the Talking Therapies service, compared to those using CBT-GSH for the first time, when taking their characteristics (like age) into account?

Participants will:

* Choose their preferred treatment
* Complete 6 sessions of either CAT-GSH or CBT-GSH
* Sessions will be weekly or bi-weekly
* Complete routine outcome measures before, during and at the end of therapy

DETAILED DESCRIPTION:
A prospective quantitative, quasi-experimental design will be used to address the primary and secondary questions. PWPs will be trained in delivering CAT-GSH. Participants will choose between CAT-GSH and CBT-GSH and be offered a six-session contact of one-to-one GSH. The Talking Therapies service already collects routine outcome measures, which will be collated and analysed.

Procedure/Intervention The Talking Therapies services routinely perform an initial assessment when someone is referred to their services. Potential participants who meet the inclusion criteria will be identified at the assessment stage.

Tameside and Glossop Talking Therapies service procedure:

The assessor will ask if there is potential interest in a study using a screening script; if the person remains interested, the participant information sheet (PIS) and the consent form will be emailed or posted. At least 48 hours will be left to allow the participant to read the information.

The principal investigator will give a follow-up phone call to answer any potential questions, ask for preference on the therapy, and complete the consent form, which will be emailed or posted back to the Talking Therapies service once completed. The completed consent form will be saved in the site's local file and a copy of the form will be sent to the participant. If the person no longer wants to participate at this stage, the service user will receive the treatment as usual.

Leeds Mental Wellbeing Service procedure:

The assessor will ask if there is potential interest in a study using a screening script; if the person remains interested, the potential participant information sheet (PIS) and the consent form will be emailed or posted. The potential participant will be given 7 days to read the information, email the Leeds service with their preferred treatment, and return the signed consent form to the service if the potential participant does not request further information. 14 days will be given if the participant asks for the material to be posted. If the potential participant requests further information, the clinical lead and principal investigator will contact the potential participant to discuss this. The completed consent form will be saved in the site's local file and a copy will be sent to the participant. If the person no longer wants to participate at this stage or has not emailed within 7 days or returned the forms by post within 14 days, the service user will receive the treatment as usual, so there are no delays.

All services procedure:

The Talking Therapies services collect routine outcome measures, demographics and other data as standard. Sessions can take place face-to-face, online, or by telephone. The sessions last 35 minutes, for a total of six sessions. Sessions are carried out weekly or bi-weekly.

The psychological wellbeing practitioner (PWP) will record the third session with the participant, so the research team can perform a randomly selected competency check on the CBT-GSH and CAT-GSH delivered to service users. The recording will be sent to the research team, with no personally identifiable information on the file name. However, due to the nature of recordings, they may contain identifiable information. Participants will be made aware of this in the PIS.

The analysis stage will aim to start in December 2025, to explore the outcome measure data.

ELIGIBILITY:
Inclusion Criteria:

* Previously received CBT-GSH at same participating NHS Talking Therapies service
* Presenting with anxiety or depression
* Deemed suitable for step 2 low-intensity therapy, through assessment by a qualified PWP

Exclusion Criteria:

* Previously received high-intensity therapy since receiving CBT-GSH
* The previous treatment episode was in another NHS Talking Therapies service.
* Not fluent in English

Individuals who are not fluent in English will be excluded from the study due to not having translated CAT-GSH workbooks available and limited funding to translate any workbooks.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Composite score (Generalised Anxiety Disorder-7 (GAD-7), Patient health Questionaire-9 (PHQ-9) and Work and Social Adjustment Scale (WSAS)) | From enrolment to the end of treatment after 6 sessions, weekly or bi-weekly. 6-12 weeks.
  Routine outcome measures, Generalised Anxiety Disorder-7 (GAD-7), Patient Health Questionaire-9 (PHQ-9) and Work and Social Adjustment Scale (WSAS) collected before, during and after treatment will be combined into composite scores.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | From enrolment to the end of treatment at 6-12 weeks. Sessions weekly or bi-weekly.
  Routine outcome measure, collected as part of normal treatment at the NHS Talking Therapy site - Patient Health Questionnaire-9 (PHQ-9). Collected before, during and after treatment. The PHQ-9 uses a 9-item scale with a total severity score of 0-27. Higher scores indicate greater depression and the clinical cut-off point indicating significant depression is ≥10.
Generalised Anxiety Disorder (GAD-7) | From enrolment to the end of treatment at 6-12 weeks. Sessions weekly or bi-weekly.
  Routine outcome measure, collected as part of normal treatment at the NHS Talking Therapy site - Generalised Anxiety Disorder-7 (GAD-7). Collected before, during and after treatment. The GAD-7 uses a 7-item scale with a total severity score ranging from 0 to 21. Higher scores indicate greater anxiety and the clinical cut-off indicating significant anxiety is ≥8

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Laphan, Principal Investigator — University of Sheffield
Locations (2):
- United Kingdom (2):
  - Tameside and Glossop NHS Talking Therapies Service, Ashton-under-Lyne
  - Leeds Mental Wellbeing Service, Leeds

IPD SHARING:
Plan to Share IPD: Yes
Only anonymized data will be shared. Personal data will not be.
Supporting Information: Study Protocol
Time Frame: At the end of the study (approximately May 2026), data will be stored on the University of Sheffield's ORDA (online research hub) for 10 years according to the University of Sheffield's retention period.
Access Criteria: Information can be requested through ORDA by those who qualify for membership.

REFERENCES:
- [Background] Williams R, Farquharson L, Palmer L, Bassett P, Clarke J, Clark DM, Crawford MJ. Patient preference in psychological treatment and associations with self-reported outcome: national cross-sectional survey in England and Wales. BMC Psychiatry. 2016 Jan 15;16:4. doi: 10.1186/s12888-015-0702-8. PMID 26768890
- [Background] Wakefield S, Delgadillo J, Kellett S, White S, Hepple J. The effectiveness of brief cognitive analytic therapy for anxiety and depression: A quasi-experimental case-control study. Br J Clin Psychol. 2021 Jun;60(2):194-211. doi: 10.1111/bjc.12278. Epub 2021 Jan 17. PMID 33458855
- [Background] Simmonds-Buckley M, Osivwemu EO, Kellett S, Taylor C. The acceptability of cognitive analytic therapy (CAT): Meta-analysis and benchmarking of treatment refusal and treatment dropout rates. Clin Psychol Rev. 2022 Aug;96:102187. doi: 10.1016/j.cpr.2022.102187. Epub 2022 Jul 18. PMID 35914380
- [Background] Owen K, Laphan A, Gee B, Lince K. Evaluating cognitive analytic therapy within a primary care psychological therapy service. Br J Clin Psychol. 2023 Sep;62(3):663-673. doi: 10.1111/bjc.12430. Epub 2023 Jun 14. PMID 37317047
- [Background] Meadows J, Kellett S. Development and Evaluation of Cognitive Analytic Guided Self-Help (CAT-SH) for Use in IAPT Services. Behav Cogn Psychother. 2017 May;45(3):266-284. doi: 10.1017/S1352465816000485. Epub 2017 Mar 22. PMID 28325165
- [Background] Lorimer B, Kellett S, Giesemann J, Lutz W, Delgadillo J. An investigation of treatment return after psychological therapy for depression and anxiety. Behav Cogn Psychother. 2024 Mar;52(2):149-162. doi: 10.1017/S1352465823000322. Epub 2023 Aug 11. PMID 37563726
- [Background] Kellett S, Simmonds-Buckley M, Limon E, Hague J, Hughes L, Stride C, Millings A. Defining the Assessment and Treatment Competencies to Deliver Low-Intensity Cognitive Behavior Therapy: A Multi-Center Validation Study. Behav Ther. 2021 Jan;52(1):15-27. doi: 10.1016/j.beth.2020.01.006. Epub 2020 May 20. PMID 33483113
- [Background] Hallam C, Simmonds-Buckley M, Kellett S, Greenhill B, Jones A. The acceptability, effectiveness, and durability of cognitive analytic therapy: Systematic review and meta-analysis. Psychol Psychother. 2021 Mar;94 Suppl 1:8-35. doi: 10.1111/papt.12286. Epub 2020 Jun 15. PMID 32543107
- [Background] Bohnke JR, Lutz W, Delgadillo J. Negative affectivity as a transdiagnostic factor in patients with common mental disorders. J Affect Disord. 2014 Sep;166:270-8. doi: 10.1016/j.jad.2014.05.023. Epub 2014 May 27. PMID 25012441
- [Background] Wray A, Kellett S, Bee C, Smithies J, Aadahl V, Simmonds-Buckley M, McElhatton C. The acceptability of cognitive analytic guided self-help in an Improving Access to Psychological Therapies service. Behav Cogn Psychother. 2022 Sep;50(5):493-507. doi: 10.1017/S1352465822000194. Epub 2022 May 16. PMID 35575218
- [Background] Kellett S, Bee C, Smithies J, Aadahl V, Simmonds-Buckley M, Power N, Dugen-Williams C, Fallon N, Delgadillo J. Cognitive-behavioural versus cognitive-analytic guided self-help for mild-to-moderate anxiety: a pragmatic, randomised patient preference trial. Br J Psychiatry. 2023 Sep;223(3):438-445. doi: 10.1192/bjp.2023.78. PMID 37395600